CLINICAL TRIAL: NCT05988541
Title: Overview of Surgically Treated Rotator Cuff Injury Patients and Rotator Cuff Integrity 5 Years After Atraumatic Rotator Cuff Tendon Repair.
Brief Title: Rotator Cuff Integrity and Clinical Outcomes 5 Years After Repair.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Tikk2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: rotator cuff injury; rotator cuff tears; sonography; shoulder injuries; atraumatic tears; shoulder pathology; shoulder ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture; Shoulder Injuries | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atraumatic rotator cuff tendon repair (Other): Ultrasonography imaging of the operated shoulder
  Interventions: Diagnostic Test: Ultrasonography imaging; Diagnostic Test: American Shoulder and Elbow Surgeons (ASES) Score; Diagnostic Test: The Constant-Murley score (CMS); Diagnostic Test: The Disabilities of the Arm, Shoulder and Hand (DASH)
- Contralateral shoulder (Other): Ultrasonography imaging of the contralateral shoulder
  Interventions: Diagnostic Test: Ultrasonography imaging; Diagnostic Test: American Shoulder and Elbow Surgeons (ASES) Score; Diagnostic Test: The Constant-Murley score (CMS); Diagnostic Test: The Disabilities of the Arm, Shoulder and Hand (DASH)

INTERVENTIONS:
Diagnostic Test: Ultrasonography imaging — Ultrasonography: rotator cuff tendons (supraspinatus, infraspinatus, subscapularis) integrity, long head of the biceps tendon integrity and location, SASD (subacromial-subdeltoid) bursitis, synovitis and muscle atrophy.
Diagnostic Test: American Shoulder and Elbow Surgeons (ASES) Score — The patient self-assessment (pASES) includes 6 pain items and 10 functional items that are shoulder specific (Angst, 2008).
  The pASES form has 3 sections: pain, instability, ADLs (Goldhahn, 2008).
  1. Pain section: 4 questions with yes/no responses, 1 question covering number of pain tablets per day, and a VAS (visual analogue scale) from 0 (no pain) to 10 (worst pain).
  2. Instability section: 2 questions (1. Response yes/no about feelings of instability, 2. Quantify instability from 0 (stable) to 10 (very unstable)).
  3. Activities of daily living (ADLs): Each shoulder is included (affected/non affected), 10 items, with a 4 point ordinal scale, range: 0 (unable to perform activity) to 3 (no difficulty in doing activity) (Goldhahn 2008).
Diagnostic Test: The Constant-Murley score (CMS) — The test is divided into four subscales: pain (15 points), activities of daily living (ADL) (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points).
Diagnostic Test: The Disabilities of the Arm, Shoulder and Hand (DASH) — 30-item self-report questionnaire designed to assess symptoms and function of the entire upper extremity.
  Total scores range from 0 (minimum) to (100) maximum.

SUMMARY:
The study gives an overview of surgically treated rotator cuff injury patients in Tartu University Hospital Sports Traumatology Centre during 2013-2019 and evaluates the integrity of rotator cuff at minimum 5 years after atraumatic rotator cuff tendon repair.

First stage of the study describes the study population, etiology of the injury (traumatic/atraumatic) and aims to answer the question whether the arthroscopic findings are in line with the preoperative imaging studies or not.

Second stage of the study focuses on atraumatic tendon tears assessing structural integrity of the tendons 5 years after repair using ultrasound imaging. The main question is - does the findings correlate with clinical outcomes and patient satisfaction.

Participants of the second phase of the study will be asked for an appointment to have their shoulders examined with ultrasonography and clinical outcomes are measured using the American Shoulder and Elbow Surgeons (ASES) Score, The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire and The Constant-Murley score (CMS).

DETAILED DESCRIPTION:
High numbers of re-tear after rotator cuff surgery have been shown, though not always influencing patient satisfaction. If there is an atraumatic tendon tear, the risk of having a contralateral rotator cuff tendon tear is high.

The aim is to study surgically treated rotator cuff injury patients 5 years after repair to evaluate tendon integrity on ultrasonography and answer the question do the findings correlate with functionality and patient satisfaction. It has been shown that people over the age of 66 who have been diagnosed with rotator cuff tendon tear, have up to 50 % chance of having a rotator cuff tendon tear in contralateral shoulder (Yamaguchi, et al. 2006). Therefore the study will evaluate the function and the integrity of the rotator cuff in both shoulders.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent rotator cuff repair by three orthopaedic surgeons at the Tartu University Hospital Sports Traumatology Centre between 2013 and 2019.
* Subject gives an informed consent and is willing to come for one outpatient visit.

Exclusion Criteria:

* Patients who underwent rotator cuff repair for traumatic tears are excluded from clinical assessment (stage II).
* Patients who underwent revision surgery are excluded from clinical assessment (stage II).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonography | 5 years after primary repair
  Integrity of the rotator cuff tendons

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) score | 5 years after primary repair
  The higher the score, the better the outcome.
Constant-Murley score (CMS) | 5 years after primary repair
  The higher the score, the higher the quality of the function.
The Disabilities of the Arm, Shoulder and Hand (DASH) | 5 years after primary repair
  The higher the score, more severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Tikk, MD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No